CLINICAL TRIAL: NCT07046026
Title: Work Design Interventions for Older Workers During Consecutive Days in the Heat
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Riana Pryor, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00112234
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Hyperthermia; Fatigue; Heat; Work-Related Condition
Keywords: hyperthermia; worker
MeSH Terms: conditions — Hyperthermia; Heat Stress Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard work pace first (Active Comparator): The order of the interventions is standard work pace first, followed by the rest trial second.
  Interventions: Behavioral: Standard work pace; Behavioral: Additional rest breaks
- Additional rest breaks first (Experimental): The order of the interventions is the additional rest breaks first and the standard work pace second.
  Interventions: Behavioral: Standard work pace; Behavioral: Additional rest breaks

INTERVENTIONS:
Behavioral: Standard work pace — On two consecutive days, participants will work at a standard pace of one box per minute during the box carrying protocol
Behavioral: Additional rest breaks — On two consecutive days, participants will work at the standard work pace during the box carrying protocol and have superimposed 5 minutes of rest every 30 minutes.

SUMMARY:
The goal of this project is to compare different ways to schedule a workday to see if older workers should follow a specific work protocol to reduce strain on the heart and muscles across two consecutive days of work.

Participants will come to the lab a total of six times. During four of the visits participants will complete a box carrying task, simulating unloading a delivery truck. This will take place in a hot and humid room to simulate being outdoors during the summer.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* 18-29 years old and 40-65 years old
* Completes at least 120 minutes of moderate to vigorous physical activity each week for at least the past 4 weeks
* Resistance trained or have recently held a job involving box carrying or a similar task

Exclusion Criteria:

* History of cardiovascular, metabolic, respiratory, neural, or renal disease
* Hypertensive (systolic blood pressure > 139 mmHg or diastolic blood pressure > 89 mmHg) or tachycardic (resting heart rate > 100 bpm) during the screening visit
* Current nicotine use or previous use within the past 6 months
* Current of previous musculoskeletal injury limiting physical activity
* A positive pregnancy test at any point during the study
* Currently breastfeeding
* Study physician discretion based on any other medical condition or medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2028-09 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Cardiac Troponin | 2 hours following work protocol, approximately 6 hours into the trial
  Serum cardiac troponin concentration
Maximum Core Temperature | End of work protocol, approximately 4 hours into the trial
  Highest core temperature attained during the work protocol

IPD SHARING:
Plan to Share IPD: Yes
A spreadsheet of the cleaned, de-identified individual data for all variables will be shared on at clinicaltrials.gov without restriction to ensure public availability. Individual data will be identified using unique participant identifier numbers. In addition to the datasets, a study protocol, data dictionary defining and describing all variables, and data collection instruments will be shared and associated with the relevant datasets.
Supporting Information: Study Protocol
Time Frame: Data from this project will be made available as soon as able and no later than the time of the final publication. Original data will be preserved indefinitely after the end of the funding period.
Access Criteria: Pooled and de-identified data will be made available to interested researchers upon email request.